CLINICAL TRIAL: NCT07160556
Title: Causes of Delayed Presentation of Patients With Myocardial Infarction to a Tertiary Care Hospital: A Cross-Sectional Study
Brief Title: Causes of Delayed Presentation of MI Patients to a Tertiary Care Hospital
Acronym: Delay-MI
Status: Completed | Type: Observational
Sponsor: Bacha Khan Medical College (Other)
Responsible Party: Principal Investigator, Malik Shayan Ali Khan, doctor, Bacha Khan Medical College
Other Study IDs: Ref no. 524 /BKMC
Record Dates: First submitted 2025-08-23; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Myocardial Infarction; DM; HTN-Hypertension
Keywords: Myocardial Infarction; Delayed presentation; Acute Coronary Syndrome; Cardiovascular Disease
MeSH Terms: conditions — Myocardial Infarction; Hypertension; Acute Coronary Syndrome; Cardiovascular Diseases | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational — no intervention was required for this cross sectional study

SUMMARY:
This study is being done to learn more about people who have had a heart attack, also called a myocardial infarction (MI). A heart attack happens when blood flow to the heart muscle is blocked, causing damage. The purpose of this study is to better understand the causes of delayed presentation and effects of the factors that caused delayed presentation.

We will collect information about patients' medical history, treatments, and recovery after their heart attack. This information may include blood tests, heart imaging, medications, and lifestyle factors. By studying these patients, we hope to find patterns that can help doctors predict complications, improve treatment, and reduce the chance of another heart attack.

The results of this study may help health care providers give better care and guidance to patients and families living with heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older with a confirmed diagnosis of myocardial infarction (STEMI or NSTEMI).
* Ability to provide informed consent (or consent from a legally authorized representative if patient is incapacitated).

Exclusion Criteria:

* Severe comorbid illness (e.g., advanced cancer, end-stage renal or liver disease) that may limit survival or affect study outcomes.
* Inability to comply with follow-up requirements (e.g., cognitive impairment, lack of contact information, or unwillingness to participate)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients diagnosed with acute myocardial infarction (MI) admitted to the cardiology department. Eligible participants include both male and female patients who meet the clinical and diagnostic criteria for MI and provide informed consent
Sampling Method: Non-Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Number and percentage of MI patients identifying specific barriers (e.g., lack of awareness, distance, transport issues) for delayed hospital presentation, using a researcher-designed structured questionnaire. | 6 months
  Data will be collected using a structured and standardized questionnaire. The questionnaire includes:
  1. Sociodemographic data: age, gender, BMI, employment status, past history of MI, and comorbidities.
  2. Knowledge of MI symptoms and severity.
  3. Pre-hospital details: first medical contact, transportation, and time to hospital.
  4. In-hospital details: time to diagnosis and treatment.
  Responses will be summarized as frequency and percentage distributions for categorical variables (e.g., gender, employment, comorbidities), and mean ± SD for continuous variables (e.g., age, BMI).

CONTACTS AND LOCATIONS:
Locations (1):
- Mardan Medical Comlex, Mardan, Mardan, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No